CLINICAL TRIAL: NCT01415297
Title: A Phase I Dose Escalation Study of NKP-1339 Administered on Days 1, 8 and 15 of Each 28-Day Cycle in Patients With Advanced Solid Tumors Refractory to Treatment
Brief Title: Dose Escalation Study of NKP-1339 to Treat Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Niiki Pharma Inc. (Industry)
Responsible Party: Sponsor
Organization: Intezyne Technologies, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NKP-1339-09-002
Record Dates: First submitted 2011-08-03; First posted 2011-08-11 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Solid Tumors
Keywords: Phase 1; advanced solid tumors
MeSH Terms: interventions — NKP-1339

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NKP-1339 (Experimental): NKP-1339 will be administered in single patient cohorts until ≥ Grade 2 toxicity encountered, at which time cohorts converted to a standard 3 + 3 dose escalation scheme.
  When MTD is reached, an expanded cohort of up to 25 patients will be enrolled at the MTD.
  Interventions: Drug: NKP-1339

INTERVENTIONS:
Drug: NKP-1339 — NKP-1339 is administered as a 30-90 minute IV infusion (based on volume to be infused) on days 1, 8, and 15 of a 28 day cycle.
  Other Names: IT-139

SUMMARY:
The purpose of this study is to determine the safety and maximal tolerated dose of NKP-1339, a ruthenium containing compound administered intravenously on a weekly schedule, in patients with advanced solid tumors. The responses to treatment in this population will be evaluated. In addition, the PD and PK properties of the compound will be explored.

DETAILED DESCRIPTION:
NKP-1339 is a novel GRP78 targeted ruthenium based anti-cancer compound which is intravenously administered. GRP78 is a key regulator of misfolded protein processing, which is unregulated in cancer cells. In nonclinical anti-tumor studies, NKP-1339 showed activity against many tumor types, including those resistant to platinum and other standard anti-cancer agents. This Phase I trial evaluates the safety, tolerability, maximum tolerated dose, pharmacokinetics, and pharmacodynamics of NKP-1339.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years with histologically or cytologically confirmed advanced solid tumors refractory to standard therapies who have signed an IRB approved Informed Consent Form (ICF).
* ECOG PS 0 or 1.
* Adequate hematologic, hepatic and renal function
* Minimum life expectancy ≥ 12 weeks

Exclusion Criteria:

* No supplemental Iron, i.e., therapeutic or as part of a multivitamin regimen.
* No chemotherapy, immunotherapy, or radiotherapy for < 4 weeks, BMTs < 9 months or major surgery < 3 weeks.
* No symptomatic central nervous system metastases. No primary brain tumors or known brain metastasis unless clinically stable and on stable or reducing dose of steroids.
* No evidence of ischemia, MI within the past 6 months, or other significant abnormality on ECG.
* No clinically significant active infection including HIV, hepatitis B, or hepatitis C.
* No Peripheral neuropathy ≥ Grade 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2012-05 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with related adverse events | 8 weeks
  The incidence and severity of related adverse events and laboratory abnormalities will be used to assess the safety and tolerability of NKP-1339.

SECONDARY OUTCOMES:
Composite of pharmacokinetics | 0, 0.25, 0.5, 1, 2, 4, 6, 10 and 24 hours
  Plasma and urine samples will be analyzed to determine Cmax, Tmax, AUC, terminal elimination rate, elimination half-life, clearance,and volume of distribution.
To report any responses to NKP-1339 in subjects with advanced tumors | >8 weeks
  Tumor assessments every 2 cycles if patients continue treatment beyond 2 Cycles. Treatment is allowed beyond 2 cycles in patients who achieved at least stable disease, at the discretion of investigator and consent of the patient.
To explore pharmacodynamic endpoints which may be of use in the further development of NKP-1339 | 8 weeks
  Transferrin, transferrin receptor and GRP-78 in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel D. Von Hoff, MD, Principal Investigator — TGEN Clinical Research Services at Scottsdale Healthcare; Howard A. Burris, III, MD, Principal Investigator — The Sarah Cannon Research Institute
Locations (2):
- United States (2):
  - TGEN Clinical Research Services at Scottsdale Healthcare, Scottsdale, Arizona
  - The Sarah Cannon Research Institute, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Burris HA, Bakewell S, Bendell JC, Infante J, Jones SF, Spigel DR, Weiss GJ, Ramanathan RK, Ogden A, Von Hoff D. Safety and activity of IT-139, a ruthenium-based compound, in patients with advanced solid tumours: a first-in-human, open-label, dose-escalation phase I study with expansion cohort. ESMO Open. 2017 Feb 23;1(6):e000154. doi: 10.1136/esmoopen-2016-000154. eCollection 2016. PMID 28848672